CLINICAL TRIAL: NCT06493565
Title: Routine Endoscopic Evaluation of Colorectal Anastomoses for Early Detection of Anastomotic Leakage (REAL-study)
Brief Title: Routine Endoscopic Evaluation of Colorectal Anastomoses for Early Detection of Anastomotic Leakage
Acronym: REAL
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Roel Hompes, MD, Dr. Roel Hompes, principal investigator, Amsterdam UMC, location VUmc
Other Study IDs: REAL-study
Record Dates: First submitted 2024-06-03; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Anastomotic Leak Rectum
Keywords: Anastomotic leakage; Colorectal cancer; Rectoscopy; Endoscopy; Point-of-care
MeSH Terms: conditions — Anastomotic Leak; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Routine endoscopic anastomosis inspection — The routine care pathway for early detection of anastomotic leakage includes:
  * C-reactive protein guided imaging
  * Rectoscopy of the anastomosis three to six days after surgery
  * Rectoscopy of the anastomosis two to three weeks after surgery

SUMMARY:
The objective of this international prospective observational study is to evaluate the implementation of a point-of-care digital rectoscope (LumenEye) into routine care to detect colorectal anastomotic leakage in the early postoperative period.

The study includes patients undergoing a colorectal resection with colorectal or coloanal anastomosis ≤15 centimeters from the anorectal junction. The participating centers consist of expert colorectal units in various countries.

The primary endpoint for the study is the time to diagnosis of anastomotic leakage.

DETAILED DESCRIPTION:
Anastomotic leakage (AL) following colorectal surgery may occur in up to 20% of patients. Treatment success for AL largely depends on its timely initiation. Relatedly, early diagnosis can avoid severe consequences such as major reoperations, oncological compromise, definitive stomas and even mortality. AL presents in a variety of clinical manifestations, ranging from faecal peritonitis with sepsis to occult or with minimal symptoms. The latter can be subject to delayed diagnosis, possibly owing to clinical pathways that are mainly focussed on signs of infection in the initial postoperative period. If left untreated, a subclinical manifestation of AL can develop into chronic pelvic sepsis. AL that progresses to this chronic stage presents a whole new set of challenges including high-risk salvage surgery with poor functional outcome, and must be avoided whenever possible. The impact of chronic AL on quality of life and the related socioeconomic burden is rarely reported, but is certainly extensive.

Endoscopic assessment of the anastomosis in the early postoperative period may prove beneficial, particularly for patients with minimal or absent clinical signs of infection. In a prospective cross-sectional study, the endoscopic evaluation of rectal anastomoses between days five and eight after surgery in 90 clinically unremarkable patients, led to the diagnosis of 11 (12.2%) additional ALs. This demonstrates that a pro-active diagnostic approach using endoscopy has the potential to mitigate delayed diagnosis of AL that manifests occult or with minimal symptoms. We hypothesized that a multicentre implementation of routine endoscopic assessment of the anastomosis in the early postoperative period can lead to a reduced time to diagnosis of AL.

The objective of this study is to evaluate the implementation of a point-of-care digital rectoscope (LumenEye) into routine care to detect colorectal anastomotic leakage in the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. The participant underwent an open or minimally invasive, sphincter preserving surgery with the construction of a colorectal or coloanal anastomosis ≤15 centimetres from the anorectal junction.
3. Adequate comprehension of the country specific or English language
4. Written informed consent

Exclusion Criteria:

1. Inability to adopt the required positioning for anorectal endoscopic examination (i.e. left lateral position)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients undergoing a colorectal resection with anastomosis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis of anastomotic leakage | 1 year

SECONDARY OUTCOMES:
Diagnostic accuracy of point-of-care rectoscopy for detection of AL | 1 year
  Determination of the sensitivity, specificity, negative- and positive predictive values for detecting AL with regards to CT-scan, flexible endoscopy and clinical findings
Patient reported comfort score for diagnostic endoscopy (Gloucester Comfort Scale), | 1 year
  a score of 1 refers to no discomfort while 5 is associated with severe discomfort
Hospital costs of the diagnostic protocol for detection of AL | 1 year
  The direct hospital costs related to the diagnostics aimed at detecting AL
Readmission rate | 1 year
Reintervention rate | 1 year
  Amount of reinterventions and specification
Mortality | 1 year
(Permanent) stoma rate at one year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roel Hompes, MD PhD, Principal Investigator — Amsterdam UMC
Locations (5):
- Bordeaux Colorectal Institute Academy, Bordeaux, France
- Humanitas Research Hospital, Milan, Italy
- Amsterdam UMC, Amsterdam, Netherlands
- University Hospital Vall D'Hebron, Barcelona, Spain
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided